CLINICAL TRIAL: NCT05146440
Title: Phase Ib/II Multicohort Trial of Different Schemes of PM14 in Monotherapy and in Combination with Radiotherapy in Soft Tissue Sarcomas and Other Solid Tumors
Brief Title: Multicohort Trial of Different Schemes of PM14 in Monotherapy and in Combination with Radiotherapy in Soft Tissue Sarcomas and Other Solid Tumor
Acronym: PRIME
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-83
Record Dates: First submitted 2021-11-12; First posted 2021-12-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Advanced Soft-tissue Sarcoma; Advanced L-sarcomas; Other Advanced Sarcomas; Advanced Solid Tumor; Localized Soft-tissue Sarcoma

STUDY DESIGN:
Intervention Model Description: Phase Ib/II, multicohort, single arm, open-label, multicenter, international clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PM14 in monotherapy and in combination with radiotherapy in STS and other solid tumors (Experimental): Cohort A : Phase I. PM14 24-h IV 21-d cycles, up to PD or toxicity. Dexamethasone recommended.
  Cohort B: Phase I. PM14 3-h IV infusion 3 d 21-d cycles, up to PD or toxicity. Dexamethasone recommended.
  Cohort E: PM14 at RP2D. Dexamethasone recommended. 21-d cycles up to PD or toxicity.
  Cohort F: PM14 at the RP2D. Dexamethasone recommended. 21-d cycles up to PD or toxicity.
  Cohort C: Phase I: PM14 at the RP2D, 21-d cycles in combination with radiotherapy, up to PD or toxicity. Dexamethasone recommended. Radiation therapy 3Gy/f 10 d. Phase II: PM14 at RP2D with radiation therapy.
  Cohort D: Phase I: PM14 at the RP2D, 3 x 21-d cycles in neoadjuvant setting, in combination with radiotherapy. Dexamethasone recommended. Radiation therapy 1.8Gy/f 25 d. Phase II: PM14 at RP2D with radiation therapy.
  Interventions: Drug: PM14

INTERVENTIONS:
Drug: PM14 — Pharmaceutical form: PM14 drug product is provided as a sterile lyophilized powder for concentrate for solution for infusion with a strength of 5.0 mg of the active moiety.
  Route of administration: PM14 drug product was developed for administration by the i.v. route. Before use, the vials are reconstituted with 10 mL of sodium chloride 9 mg/mL (0.9%) solution for infusion to give a solution containing 0.5 mg/mL of PM14. Prior to administration, the reconstituted DP solution should be further diluted with sodium chloride 9 mg/mL (0.9%) solution for infusion. Each vial of PM14 5.0 mg is a single use vial.

SUMMARY:
Phase Ib/II, multicohort, single arm, open-label, multicenter, international clinical trial, with 6 cohorts (advanced STS, advanced L-sarcomas, other advanced sarcomas, advanced solid tumors, and localized STS) with 4 sites in Spain for phase I.

The aim of this study is to explore different infusions of PM14 (longer or repeated) in order to obtain a potentially better efficacy and similar toxicity profile in advanced soft tissue sarcoma patients as monotherapy and also in other solid tumors as concomitant treatment with radiation therapy.

Treatment

Cohort A

A phase I dose-finding stage for PM14 is planned with an estimated number of 20-25 patients. PM14 will be tested at different dose levels in 24-h IV infusion on day 1 of 21-day cycles, up to progression or unacceptable toxicity. Premedication with dexamethasone is recommended on the day before treatment initiation.

Cohort B

A phase I dose-finding stage for PM14 is planned with an estimated number of 20-25 patients. PM14 will be tested at different dose levels in 3-h IV infusion during 3 consecutive days (days 1-3) of 21-day cycles, up to progression or unacceptable toxicity. Premedication with dexamethasone is recommended on the day before treatment initiation.

Cohort E

PM14 will be administered at the recommended phase II dose (RP2D) according to the most convenient scheme. Cycles will be administered by central venous port. Premedication with dexamethasone is recommended on the day before treatment initiation. Cycles will be repeated every 21 days up to progression or unacceptable toxicity.

Cohort F

PM14 will be administered at the RP2D according to the most convenient scheme. Cycles will be administered by central venous port. Premedication with dexamethasone is recommended on the day before treatment initiation. Cycles will be repeated every 21 days up to progression or unacceptable toxicity.

Cohort C

Phase I: PM14 will be administered at the RP2D according to the most convenient scheme in 21-day cycles, at at different dose levels in combination with radiotherapy, up to progression or unacceptable toxicity. Cycles will be administered by central venous port. Premedication with dexamethasone is recommended on the day before treatment initiation and during 2 additional days (in the 24-hour infusion) and during 3 additional days (in the 3-hour infusion). Radiation therapy will start within 1 hour of PM14 infuser disconnection and will be administered with 3 Gy per fraction for 10 days (30 Gy in total).

Phase II: PM14 will be administered at RP2D concomitant with radiation therapy.

Cohort D

Phase I: PM14 will be administered at the RP2D according to the most convenient scheme, in up to 3 x 21-day cycles in neoadjuvant setting, at different dose levels in combination with radiotherapy. Cycles will be administered by central venous port. Premedication with dexamethasone is recommended on the day before treatment initiation. Radiation therapy will start within 1 hour of PM14 infuser disconnection and will be administered with 1.8 Gy per fraction for 25 days (45 Gy in total).

Phase II: PM14 will be administered at RP2D concomitant with radiation therapy.

DETAILED DESCRIPTION:
Cohort A and B (Phase I, PM14 monotherapy, advanced STS): 20-25 patients approximately per cohort.

Cohort E (Phase II, PM14 monotherapy, advanced L-sarcomas): 28 patients; (Simon's two-stage Minimax design), errors: α= 0.05; β=0.80, option related to efficacy = 35% (6-month PFSR) (Sample size 15+13), success in 6-month PFSR of ≤ 15% will be considered as unacceptable (H0), and would not warrant further investigation (null hypothesis). Success in 6-month PFSR of ≥ 35% will be considered as an acceptable result warranting further investigation of the investigational drug (H1, alternative hypothesis). A total of 15 eligible and treated patients will be included in the first stage of the study. If ≤ 2 successes are observed, the trial will be stopped in this cohort with the conclusion that the experimental treatment should not be further investigated. Else (≥ 3 successes), patients will continue to be accrued until 28 eligible patients enter the study. If 8 or more successes are observed in those 28 patients, it will be concluded that the results of this trial warrant further investigation.

Cohort F (Phase II, PM14 monotherapy, other advanced sarcomas): 29 patients; (Simon's two-stage Optimal design), errors: α= 0.05; β=0.80. option related to efficacy = 30% (6-month PFSR) (Sample size 10+19), success in 6-month PFSR of ≤ 10% will be considered as unacceptable (H0), and would not warrant further investigation (null hypothesis). Success in 6-month PFSR of ≥ 30% will be considered as an acceptable result warranting further investigation of the investigational drug (H1, alternative hypothesis). A total of 10 eligible and treated patients will be included in the first stage of the study. If ≤ 1 successes are observed, the trial will be stopped in this cohort with the conclusion that the experimental treatment should not be further investigated. Else (≥ 2 successes), patients will continue to be accrued until 29 eligible patients enter the study. If 6 or more successes are observed in those 29 patients, it will be concluded that the results of this trial warrant further investigation.

Cohort C (Best scheme of PM14 plus RTP in advanced sarcoma, head & neck, other solid tumors)

Phase I (advanced): pulmonary and/or abdominal cohort (2 dose levels), head and neck cohort (2dose levels). 25 patients approximately.

Phase II (advanced STS): errors: α=0.05; β=0.80, option related to efficacy = 50% (ORR in irradiated nodules) (Sample size 9+15), success in ORR of ≤ 25 % will be considered as unacceptable (H0), and would not warrant further investigation (null hypothesis). Success in ORR of ≥ 50% will be considered as an acceptable result warranting further investigation of the investigational drug (H1, alternative hypothesis). A total of 9 eligible and treated patients will be included in the first stage of the study. If ≤ 2 successes are observed, the trial will be stopped in this cohort with the conclusion that the investigational combination should not be further investigated. Else (≥ 3 successes), patients will continue to be accrued until 24 eligible patients enter the study. If 10 or more successes are observed in those 24 patients, it will be concluded that the results of this trial warrant further investigation.

Cohort D (Best scheme of PM14 plus RTP in localized intermediate sarcoma)

Phase I (localized sarcoma): 2 dose levels, 10 patients approximate ly. Phase II (localized "intermediate risk" STS): errors: α=0.05; β=0.80, option related to efficacy = 30% (ORR in irradiated nodules) (Sample size 10+19), success in ORR of ≤ 10% will be considered as unacceptable (H0), and would not warrant further investigation (null hypothesis). Success in ORR of ≥ 30% will be considered as an acceptable result warranting further investigation of the investigational drug (H1, alternative hypothesis). A total of 10 eligible and treated patients will be included in the first stage of the study. If ≤ 1 successes are observed, the trial will be stopped in this cohort with the conclusion that the investigational combination should not be further investigated. Else (≥ 2 successes), patients will continue to be accrued until 29 eligible patients enter the study. If 6 or more successes are observed in those 29 patients, it will be concluded that the results of this trial warrant further investigation.

ELIGIBILITY:
Inclusion Criteria:

Cohorts A, B, E, and F

1. The patient must voluntarily sign the informed consent before any study test is conducted that is not part of routine patient care.
2. Age: 18-75 years.
3. Patients must have a diagnosis of soft tissue sarcoma with metastasis, and not suitable for metastasectomy or surgery resection or not oncologically recommended metastasectomy. A centralized diagnosis confirmation will be performed and the tumor sample must be available and sent prior to inclusion to this end.
4. A centralized diagnosis of DD liposarcoma or mixoid/hypercellular liposarcoma or leiomyosarcoma must be confirmed for patients in cohort E.
5. A centralized diagnosis of other sarcomas includes: undifferentiated pleomorphic sarcoma (UPS), myxofibrosarcoma, synovial sarcoma, malignant peripheral nerve sheath tumors, sarcoma NOS, fibrosarcoma, pleomorphic rhabdomyosarcoma, pleomorphic liposarcoma, epithelioid sarcoma, clear cell sarcoma, dedifferentiated or aggressive features in solitary fibrous tumor, extraskeletal myxoid chondrosarcoma, angiosarcoma, epithelioid hemangioendothelioma,
6. Patients must have received a previous chemotherapy line in advanced disease unless contraindicated or not indicated.
7. Radiological disease progression must be documented within 6 months prior to study entry.
8. The patient must have been considered eligible for systemic chemotherapy. A maximum of two previous lines for advanced/metastatic disease are allowed.
9. Measurable disease according to RECIST v1.1 criteria.
10. Performance status ≤1 (ECOG).
11. Adequate bone marrow function (hemoglobin >10 g/dL, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3). Patients with creatinine clearance ≥ 30 mL/min (Cockcroft and Gault's formula), transaminases ≤ 3.0 times the ULN, total bilirubin ≤ ULN, are acceptable.
12. Men or women of childbearing potential must be using an effective method of contraception before entry into the study and throughout the same and for 3 months (men) and 6 months (women) after ending study treatment. Women of childbearing potential must have a negative serum or urine pregnancy test before study entry.
13. Normal cardiac function with a LVEF ≥ 50% by echocardiogram or MUGA.
14. HBV and HCV serologies must be performed prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study).
15. Patient must have a central venous catheter for PM14 treatment.

Cohort C

1. The patient must voluntarily sign the informed consent before any study test is conducted that is not part of routine patient care.
2. Age: 18-75 years.
3. Patients must have a diagnosis of advanced soft tissue sarcoma, or recurrent head & neck suitable for reirradiation or other advanced or metastatic solid tumor not suitable for metastasectomy or surgery resection or not oncologically recommended metastasectomy. A centralized diagnosis will be performed and the tumor sample must be available and sent prior to inclusion to this end. For phase II part, onlysoft tissue sarcomas will be enrolled.
4. Patients must have received a previous chemotherapy line in advanced disease.
5. Disease distribution must allow meeting with normal tissue constrains of radiation therapy. Radiation oncologist must confirm this point at local sites.
6. Metastatic spread could be present in several organs (i.e. lungs and pelvic fossa) however, not all the locations have to be irradiated.
7. Those lesions considered for radiation therapy have to be related to symptoms (for phase II).
8. It is allowed that not all the lesions will be under radiation fields. As a general rule, the priority is to select, as target-irradiating lesions, those with greater increase in size and those largest lesions if related with symptoms. Irradiating pulmonary lesions with infiltration of pleural serosa is discouraged.
9. Radiological disease progression must be documented within 6 months prior to study entry.
10. The patient must have been considered eligible for systemic chemotherapy. A maximum of two previous lines for advanced/metastatic disease are allowed.
11. The following histological subtypes can be included for the phase II part (central pathology review is mandatory before accrual): undifferentiated pleomorphic sarcoma (UPS), leiomyosarcoma, angiosarcoma, epithelial hemangioendothelioma, liposarcoma and its variants (well differentiated, dedifferentiated, myxoid/round cell, pleomorphic), synovial sarcoma, fibrosarcoma and its variants (epithelial fibrosarcoma/low grade fibromyxoid sarcoma), solitary fibrous tumor, malignant peripheral nerve sheath tumor (MPNST), myxofibrosarcoma, epithelioid sarcoma and (NOS) unclassified sarcoma.
12. Measurable disease according to RECIST v1.1 criteria.
13. Performance status ≤1 (ECOG).
14. Adequate respiratory functions: FEV1 > 1L; DLco > 40% (patients with pulmonary target lesions).
15. Adequate bone marrow function (hemoglobin > 10 g/dL, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3). Patients withcreatinine clearance ≥ 30 mL/min (Cockcroft and Gault's formula), transaminases ≤ 2.5 times the ULN, total bilirubin ≤ ULN are acceptable.
16. Men or women of childbearing potential must be using an effective method of contraception before entry into the study and throughout the same and for 3 months (men) and 6 months (women) after ending study treatment. Women of childbearing potential must have a negative serum or urine pregnancy test before study entry.
17. Normal cardiac function with a LVEF ≥ 50% by echocardiogram or MUGA.
18. HBV and HCV serologies must be performed prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study).
19. Patient must have a central venous catheter for PM14 treatment.

Cohort D

1. The patient must voluntarily sign the informed consent before any study test is conducted that is not part of routine patient care.
2. Age: 18-75 years.
3. Patients must have a diagnosis of localized soft tissue sarcoma that lacks one or more of the following risk criteria: G3, deep and > 5 cm. At least G2 is required (i.e. G3, superficial and > 5 cm; or G3 < 5 cm deep; or G2, deep and > 5 cm, etc.).
4. Patients must be diagnosed by core-biopsy and the elapsed time between biopsy and enrollment must be shorter than 6 weeks.
5. Patients must be diagnosed by central pathology review with one of the following subtypes: leiomyosarcoma, undifferentiated pleomorphic sarcoma (UPS), myxofibrosarcoma, synovial sarcoma, sarcoma NOS, fibrosarcoma, myxoid liposarcoma,dedifferentiated liposarcoma, solitary fibrous tumor (the formerly malignant subtype).
6. Only those sarcomas of limbs or trunk wall will be eligible for this cohort.
7. Disease distribution allows meeting with normal tissue constraints of radiation therapy. Radiation oncologist must confirm this point at local sites.
8. Patients must have resectable primary tumor while it is allowed to enroll patients with metastatic spread that could be potentially resectable.
9. Patients must have criteria of operability for the primary tumor.
10. The patient must have been considered eligible for systemic chemotherapy.
11. Measurable disease according to RECIST v1.1 criteria.
12. Patients have to be candidates for MRI test.
13. Performance status ≤ 1 (ECOG).
14. Adequate bone marrow function (hemoglobin > 10 g/dL, neutrophils ≥ 1,500/mm3, platelets ≥ 100,000/mm3). Patients withcreatinine clearance ≥ 30 mL/min (Cockcroft and Gault's formula), transaminases ≤ 2.5 times the ULN, total bilirubin ≤ ULN are acceptable.
15. Men or women of childbearing potential must be using an effective method of contraception before entry into the study and throughout the same and for 3 months (men) and 6 months (women) after ending study treatment. Women of childbearing potential must have a negative serum or urine pregnancy test before study entry.
16. Normal cardiac function with a LVEF ≥ 50% by echocardiogram or MUGA.
17. It should be performed HBV and HCV serologies prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study).
18. Patient must have a central venous catheter for treatment with PM14.

Exclusion Criteria:

Cohorts A, B, E, and F

1. Performance status ≥ 2 (ECOG).
2. Plasma bilirubin > ULN.
3. Creatinine > 1.6 mg/dL.
4. History of other cancer with less than 5 years free of disease with the exception of adequately treated basal cell carcinoma or in situ cervical cancer.
5. Patients who do not provide consent for mandatory biological samples (including those required for the translational study) cannot participate in the study.
6. Significant cardiovascular disease (for example, dyspnea > 2 NYHA).
7. Significant systemic diseases grade 3 or higher on the NCI-CTCAE v5.0 scale, that limit patient availability, or according to investigator judgment may significantly contribute to treatment toxicity.
8. Uncontrolled bacterial, mycotic or viral infections.
9. Women who are pregnant or breastfeeding.
10. Psychological, family, social or geographic circumstances that limit the patients' ability to comply with the protocol or informed consent.
11. Patients participating in another clinical trial or receiving any other investigational product.
12. Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion.
13. Histologies other than those described in the inclusion criteria.

Cohort C

1. Previous treatment with radiotherapy (except if previous radiotherapy treatment plus planned study radiotherapy treatment allow tissue constrains).
2. Performance status ≥ 2 (ECOG).
3. Plasma bilirubin > ULN.
4. Creatinine > 1.6 mg/dL.
5. History of other cancer with less than 5 years free of disease with the exception ofadequately treated basal cell carcinoma or in situ cervical cancer.
6. Severe COPD or other severe pulmonary diseases.
7. Significant cardiovascular disease (for example, dyspnea > 2 NYHA).
8. Significant systemic diseases grade 3 or higher on the NCI-CTCAE v5.0 scale, that limit patient availability, or according to investigator judgment may significantly contribute to treatment toxicity.
9. Patients who do not provide consent for mandatory biological samples (including those required for the translational study) cannot participate in the study.
10. Uncontrolled bacterial, mycotic or viral infections.
11. Women who are pregnant or breastfeeding.
12. Psychological, family, social or geographic circumstances that limit the patients' ability to comply with the protocol or informed consent.
13. Patients participating in another clinical trial or receiving any other investigational product.
14. Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion.
15. Histologies other than those described in inclusion criteria.

Cohort D

1. High-risk localized patients are not allowed to be enrolled (those G3, deep, and larger than 5 cm or those with risk of death at least 40% by sarculator nomogram).
2. Previous treatment with radiotherapy.
3. Primary tumor location other than those indicated in the inclusion criteria.
4. Histological subtypes other than those indicated in the inclusion criteria.
5. Unresectable or inoperable primary tumor.
6. Patients who do not provide consent for mandatory biological samples (including those required for the translational study) cannot participate in the study.
7. Performance status ≥ 2 (ECOG).
8. Plasma bilirubin > ULN.
9. Creatinine > 1.6 mg/dL.
10. History of other cancer with less than 5 years free of disease with the exception of adequately treated basal cell carcinoma or in situ cervical cancer.
11. Significant cardiovascular disease (for example, dyspnea > 2 NYHA).
12. Significant systemic diseases grade 3 or higher on the NCI-CTCAE v5.0 scale, that limit patient availability, or according to investigator judgment may significantly contribute to treatment toxicity.
13. Uncontrolled bacterial, mycotic or viral infections.
14. Women who are pregnant or breastfeeding.
15. Psychological, family, social or geographic circumstances that limit the patients' ability to comply with the protocol or informed consent.
16. Patients participating in another clinical trial or receiving any other investigational product.
17. Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Cohorts A, B, C To determine the maximum tolerated dose (MTD) of PM14 to be used as recommended phase 2 dose (RP2D). | 1 year
  The MTD will be determined by assessing adverse events according to CTCAE v5.0 and they will be used as a rule for escalating or diminishing dose levels according to the dose-limiting toxicities detailed in the protocol.
Cohorts E and F To evaluate the progression-free survival rate (PFSR) at 6 months. | 6 months
  PFSR-6m (according to central radiology review): Efficacy measured by the PFSR at 6 months, which is defined as the percentage of patients whodid not experience radiological progression according to RECIST v1.1 or death due to any cause since the date of enrollment until month 6 after date of enrollment
Cohort C phase I To determine the maximum tolerated dose (MTD) of PM14 to be used as recommended phase 2 dose (RP2D). | 1 year
  The MTD will be determined by assessing adverse events according to CTCAE v5.0 and they will be used as a rule for escalating or diminishing dose levels according to the dose-limiting toxicities detailed in the pro
Cohort C phase II To evaluate the overall response rate (ORR) in irradiated nodules only. | 8 weeks
  This objective is considered as a surrogate of palliative relief. Overall response rate (ORR) (according to central radiology review): Efficacy measured by ORR, which is defined as the number of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of response evaluable patients (according to RECIST v1.1). Only nodules included in the radiation field will be considered.
Cohort D phase I To determine the maximum tolerated dose (MTD) of PM14 to be used as recommended phase 2 dose (RP2D). | 1 year
  The MTD will be determined by assessing adverse events according to CTCAE v5.0 and they will be used as a rule for escalating or diminishing dose levels according to the dose-limiting toxicities detailed in the protocol.
Cohort D phase II To evaluate the overall response rate (ORR). | 63 days
  Overall response rate (ORR) (according to central radiology review): Efficacy measured by ORR, which is defined as the number of patients with a best overall response (BOR) of complete response(CR)or partial response (PR) divided by the number of response evaluable patients (according to RECIST v1.1).

SECONDARY OUTCOMES:
Cohorts A, B, E, F, C, D To evaluate the safety profile | 21 days
  Toxicity will be assessed by adverse events related to study drugs, detected through physical examinations and laboratory tests, and graded according to CTCAE v5.0.
Cohorts A, B, E, F, C, D To evaluate the overall response rate (ORR). | 8 weeks
  Overall response rate (ORR) (according to central radiology review): Efficacy measured by ORR, which is defined as the number of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) divided by the number of responseevaluable patients (according to RECIST v1.1).
Cohorts A, B, C, D To evaluate the median of progression-free survival (mPFS). | 8 weeks
  mPFS (according to central radiology review): Efficacy measured by mPFS, which is defined as the median of time in months from date of enrollment to date of radiological progression according to RECIST v1.1 or to date of death due to any cause, whatever occurs first.
Cohorts A, B, E, F, C To evaluate quality of life. | 3 weeks
  Quality of life: Assessed by using the European Organization for Cancer Research and Treatment quality of life questionnaire (EORTC QLQ-C30).
  For the completion of the QLQ-C30 questionnaire, values between 1 and 4 (1: not at all, 2: a little, 3: quite a bit, 4: very much) are assigned according to the patient's responses to the item, only in items 29 and 30 are They evaluate with a score of 1 to 7 (1: very poor, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, which determines the level of impact of the cancer on the patient on each of the scales. High values on the global health and function status scales indicate a better quality of life (QoL), while on the symptom scale it would indicate a decrease in QoL since it indicates the presence of symptoms associated with cancer.
Cohorts A, B, E, F, C, D To contribute to translational studies. | 4 years
  The clinical study will provide tumor and blood samples for the translational research program.
Cohorts A and B To characterize the PK of PM14 in the explored regimens. | 1 year
  The clinical study will provide blood samples for the measurement of PM14 concentration and baseline α-1-acid glycoprotein (AAG) levels.
Cohorts E, F, C To evaluate the median of overall survival (mOS). | 3 months
  mOS: Efficacy measured by mOS, which is defined as the median of time in months from dateof enrollment to date of death due to any cause.
Cohort C phase II To evaluate variations in pain. | 3 weeks
  Changes in pain: Variations in pain will be measured by the Brief Pain Inventory - Short Form (BPI-SF).
Cohort C phase II To evaluate variations in analgesic use. | 3 weeks
  Changes in analgesic use: Variations in analgesic use will be measured by the Analgesic Quantification Algorithm (AQA).
Cohort C phase II To evaluate the time to progression (TTP) of the irradiated nodules. | 3 weeks
  Time to progression (TTP) of irradiated nodules (according to central radiology review): TTP is defined as the time in months between the date of enrollment and the date of progression of irradiated nodules (not including deaths) (according to RECIST v1.1 criteria).
Cohort C phase II To evaluate the progression-free survival rate (PFSR) at 6 months. | 6 months
  PFSR-6m (according to central radiology review): Efficacy measured by the PFSR at 6 months, which is defined as the percentage of patients whodid not experience radiological progression according to RECIST v1.1 or death due to any cause since the date of enrollment until month 6 after date of enrollment.
Cohort C phase II, D To evaluate the pathological response. | 8 weeks
  Pathological response: Assessed using a predefined surgical specimen pathology form and method describing the precise percentage of tumor non-viable histological changes (hyalinosis, necrosis, cyst, differentiation etc) and percentage of viable tumor.
Cohort D phase II To evaluate relapse-free survival (RFS) at 3 years. | 3 years
  Relapse-free survival (RFS) at 3 years: Efficacy measured by RFS at 3 years, which is defined as the percentage of patients who did not experience relapse since date of surgery until year 3 after date of surgery.
Cohort D phase II To evaluate changes in MRI diffusion/perfusion parameters (exploratory). | 63 days
  MRI imaging will be evaluated to assess variations in diffusion/perfusion parameters (exploratory)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín Broto, Study Director — Hospital Universitario Fundación Jiménez Díaz; Javier Martínez Trufero, Principal Investigator — Hospital Miguel Servet; Ana Sebio, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Claudia Valverde, Principal Investigator — Hospital Vall d'Hebron
Locations (4):
- Spain (4):
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No